CLINICAL TRIAL: NCT02452489
Title: Scheme Optimization of Acupoints Compatibility and Influence Factors of the Effect
Brief Title: Different Acupoints Compatibility Difference of the Effect of Treatment of the Diabetic Gastroparesis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changchun University of Chinese Medicine (Other)
Collaborators: The First Affiliated Hospital of Hunan University of Traditional Chinese Medicine (Other); Hengyang Traditional Chinese Medicine Hospital (Other); Second People's Hospital of Hunan (Other); Jilin University (Other); Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Tie Li, 973 project management deputy director of the office, Changchun University of Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ChangchunUCM02
Record Dates: First submitted 2015-05-20; First posted 2015-05-22 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Diabetic Gastroparesis
Keywords: Different acupoints compatibility
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Single point group (Zhongwan) (Other): Patients will be acupuncture with Zhongwan(RN12).
  Interventions: Device: acupuncture
- Combination of He-Mu points group (Other): Patients in Combination of He-Mu points group,will be acupuncture with Zusanli(ST36) and Zhongwan(RN12).
  Interventions: Device: acupuncture
- Control group (Other): Patients in Control group,will be acupuncture with at the junction of deltoid and biceps.
  Interventions: Device: acupuncture

INTERVENTIONS:
Device: acupuncture — Patients will be acupuncture with Zhongwan(RN12),needle 1 times a day,30 min/time,5 days for a period of treatment,the treatment interval for two days,three intervention treatment,follow-up after 4 weeks.
  Arms: Single point group (Zhongwan)
Device: acupuncture — Patients in Combination of He-Mu points group,will be acupuncture with Zusanli(ST36) and Zhongwan(RN12),needle 1 times a day,30 min/time,5 days for a period of treatment,the treatment interval for two days,three intervention treatment, follow-up after 4 weeks.
  Arms: Combination of He-Mu points group
Device: acupuncture — Patients in Control group,will be acupuncture with at the junction of deltoid and biceps,needle 1 times a day,30 min/time,5 days for a period of treatment,the treatment interval for two days,three intervention treatment,follow-up after 4 weeks.
  Arms: Control group

SUMMARY:
With Diabetic gastroparesis as the research object, by the method of multi-center RCT and single cavity and different acupuncture acupoints compatibility treatment of diabetic gastroparesis, the inspection of gastric emptying, gastric dynamic inspection, such as validity checking means, for single cavity with different acupoints compatibility evaluate clinical efficacy of treatment of diabetic gastroparesis.

DETAILED DESCRIPTION:
In order to establish a spectrum of acupoints compatibility of the law, is clear about the factors affecting the compatibility effect of acupoints, the formation of strong operability of acupoints compatibility optimization evaluation method, the project choice of the clinical acupuncture and moxibustion have curative effect of diabetic gastroparesis as the breakthrough point of the study, carried out clinical multi-center RCT research, through objective and scientific evaluation method, comparing the effect of different acupoints compatibility.

Diabetic gastroparesis in clinical common disease, frequently-occurring disease, acupuncture curative effect is distinct, disease diagnosis, curative effect evaluation standard. Previous clinical data also show that the diabetic gastroparesis is acupuncture clinical diseases. This project by diabetic gastroparesis as the research object, research to better guide clinical practice, improve the clinical curative effect, promote acupuncture of the inheritance and innovation, promote scientification of acupuncture and moxibustion, modernization and internationalization, and will have broad prospect of application and significant scientific research value.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Diabetic Gastroparesis;
* Aged 18-60 (including 18 and 60);
* Fasting venous blood sugar ≤7.8mmol/L,2-hour post-meal blood glucose ≤ 13.6mmol/ L;
* Diabetes more than 3 years;
* Diet and exercise therapy or diet movement and exercise therapy based on the use of hypoglycemic drugs (except alpha glycosidase inhibitor) treatment, dose stable at least more than 3 months;
* Rounding out the top three months did not participate in any clinical subjects;
* Sign the informed consent and voluntary to participate in the study.

Exclusion Criteria:

* Patients with reflux esophagitis;
* Postoperative gastroparesis patients;
* Ketoacidosis, non ketosis acute complications such as hypertonic coma;
* Patients with acute cardiovascular disease, with severe trauma or surgery, severe infections, pregnancy or breast-feeding women;
* Patients with myocardial infa,acute coronary syndrome (ACS),coronary revascularization;
* Patients with severe liver disease, or the AST and/or ALT 2 times higher than normal ceiling;
* Patients with Serum creatinine kidney damage, more than 140 umol/L;
* Patients with obvious blood system diseases (either in person are not to be included in the item: Hb: men < 110 g/L, women < 100 g/L, the WBC < 3.5×109/L/L, PLT < 80×109/L);
* Patients's systolic pressure≥180mmHg,Patients's diastolic pressure≥100mmHg;
* Patients with Advanced malignant tumor or other serious wasting disease, infection and bleeding;
* Endoscopy has the organic lesion such as peptic ulcer;
* Disorders or do not fit the person and the growing experiment condition or severe complications;
* Nearly four weeks of alpha glycosidase inhibitor drugs.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Gastroparesis Symptoms Rating Scale(GCSI) | 8 weeks

SECONDARY OUTCOMES:
FBG(fasting blood-glucose) | 8 weeks
PPG(postprandial blood sugar) | 8 weeks
Gastric emptying check by Color ultrasonography | 8 weeks
Gastric emptying check by X rays | 8 weeks
Short form 36 health survey(SF-36) | 8 weeks
Self-rating anxiety scale(SAS) | 1 week
Self-Rating Depression Scale(SDS) | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Fuchun Wang, master, Study Chair — Director
Locations (1):
- The Affiliated Hospital To Changchun University of Chinese Medicine, Changchun, Jilin, China

REFERENCES:
- [Derived] Liu R, He M, Zhao X, Sun M, Cao J, Wang X, Wang X, Zhao S, Wang F, Li T. Effects of stimulating single acupoint and combination acupoints on diabetic gastroparesis: A randomised controlled trial study. J Tradit Complement Med. 2024 Jan 23;14(4):446-455. doi: 10.1016/j.jtcme.2024.01.008. eCollection 2024 Jul. PMID 39035685